CLINICAL TRIAL: NCT01404858
Title: The Impact of Lifestyle Behavior on in Vitro Fertilization (IVF) Outcome
Status: Completed | Type: Observational
Sponsor: Boston IVF (Other)
Responsible Party: Principal Investigator, Alice D. Domar, PhD, Alice D. Domar, PhD, Boston IVF
Other Study IDs: DC2011
Record Dates: First submitted 2011-07-27; First posted 2011-07-28 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-02

CONDITIONS: Infertility
Keywords: IVF; Lifestyle habits
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients undergoing IVF
  Interventions: Behavioral: There is no intervention; this is a survey only study

INTERVENTIONS:
Behavioral: There is no intervention; this is a survey only study — There is no intervention; this is a survey only study

SUMMARY:
The purpose of this study is to prospectively examine the impact of various lifestyle habits in both men and women on the outcome of in vitro fertilization. There are 25 infertility centers in the United States which use the electronic medical record collection entity eIVF, made by Practice Highway, to collect medical and demographic information on the patients who are undergoing treatment at these centers. Information on every aspect of each cycle is also electronically collected daily during each cycle. Demographic and lifestyle information will be collected on all patients prior to cycle start and lifestyle habit information will be collected each time a patient logs onto the patient portal, which averages every few days.

ELIGIBILITY:
Inclusion Criteria:

Eligible patients include, any patient whose:

* infertility clinic uses eIVF
* is scheduled to undergo an IVF cycle
* has access to the internet on a daily basis
* can read and understand English
* logs onto the patient portal on eIVF

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Men and women undergoing IVF at a infertility clinic who uses eIVF, an electronic medical record collection entity specifically for IVF patients
Sampling Method: Non-Probability Sample
Enrollment: 12800 (Actual)
Dates: Start 2011-09; Primary Completion 2014-02 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Clinical Pregnancy Rates | Approximately 28 days (1 IVF cycle)

CONTACTS AND LOCATIONS:
Overall Officials: Alice D Domar, PhD, Principal Investigator — Boston IVF
Locations (1):
- Boston IVF, Waltham, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No